CLINICAL TRIAL: NCT05852730
Title: Optimizing the Combination of Intranasal Scopolamine and Sensory Augmentation to Mitigate G-transition Induced Motion Sickness and Enhance Sensorimotor Performance. Motion Sickness Countermeasures Field Test
Brief Title: Combination of Intranasal Scopolamine and Sensory Augmentation to Mitigate G-transition Induced Motion Sickness and Enhance Sensorimotor Performance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NASA 0354 (Aim 2)
Record Dates: First submitted 2023-04-17; First posted 2023-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Motion Sickness, Space; Motion Simulation; Parabolic Flight
Keywords: Astronauts; centrifugation; parabolic; operational
MeSH Terms: conditions — Space Motion Sickness | interventions — Scopolamine; Promethazine; Meclizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DPI-386 Nasal Gel (Experimental): DPI-386 Nasal Gel, 0.4 mg
  Interventions: Drug: DPI-386 Nasal Gel
- Control (Experimental): Another form of preventative or treatment medication for motion sickness (e.g., promethazine or meclizine)
  Interventions: Drug: Other (e.g., promethazine, meclizine)

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — Subjects will self-administer DPI-386 Nasal Gel
  Other Names: scopolamine
  Arms: DPI-386 Nasal Gel
Drug: Other (e.g., promethazine, meclizine) — Subjects will self-administer other medications as available.
  Arms: Control

SUMMARY:
The primary specific aim of this Field Test aim is to evaluate the feasibility and efficacy of administering the intranasal scopolamine gel in operational field settings using both astronaut and ground-control subjects that are exposed to provocative motion as part of their assigned duties. For the ground-control subjects, these may include motion simulations (e.g., centrifuge), parabolic flights and/or Orion capsule recovery operations. Astronaut participants may choose to test Inscop during provocative preflight training exercises (e.g., centrifugation), and can choose to take the medication prophylactically to prevent symptoms or after symptom onset to treat motion sickness during the launch and/or landing mission phases. Both ground-control and astronaut participants will be required to test the medication during a training session to monitor for adverse side effects. Participants in the field test aim will complete short debrief questionnaires to capture motion sickness symptoms, side effects, and feasibility comments. The investigators will also include field "control" subjects who did not take (INSCOP) to comment on what countermeasures subjects used and their effectiveness. The investigators will be recruiting astronaut participants from free-flier missions (e.g., SpaceX Polaris Dawn), Private Astronaut Missions (e.g., Axiom), and standard missions to the International Space Station.

DETAILED DESCRIPTION:
The primary specific aim is to evaluate the use of intranasal scopolamine gel (DPI-386) in operational field settings. Both astronauts and non-astronaut participants in the field testing will be recruited to test the feasibility and efficacy of the intranasal scopolamine gel (0.4 mg dosage). This testing will include only the active drug (no placebo); however, control astronaut subjects will also be recruited who choose other motion sickness countermeasures. The goal is to recruit astronauts from free-flier missions like SpaceX Polaris Dawn (8 active, 8 control), from Private Astronaut Missions to the International Space Station (ISS) like Axiom (8 active, 8 control), and from standard missions to the International Space Station (8 active, 8 control). Astronaut participants who choose to take intranasal scopolamine gel will be required to complete a 15 min training session to learn how to apply the medication, and then a 15 min debrief on any symptoms, side effects and comments on the efficacy and feasibility of self-administering the medication. Astronaut participants will also have the option to self-administer the drug during preflight activities that involve exposure to a motion environment (e.g., centrifuge training). For each time subjects choose to self-administer the drug, subjects will be asked to complete a short 15 min survey to describe the operational environment (e.g., centrifuge levels), any symptoms subjects experienced, side effects and comment s on the efficacy and feasibility of self-administering the medication. All astronauts, both active and control, will be tasked to complete a short inflight and postflight survey (15-30 min each) to summarize symptoms by day, record what medications were taken, rate their effectiveness, and summarize their recommendations on what others can do (or avoid) to improve recovery.

This test may also involve non-astronaut test personnel during operational activities that involve provocative motion, e.g., capsule recovery simulations, centrifuge training, and parabolic flights. Participants for this part of the study will be recruited from personnel who are already involved and medically cleared for these operational activities and are interested in trying the drug to prevent or treat symptoms in addition to their primary task(s). In order to participate in these field test activities, subjects will be required to complete a 15 min training session to learn how to apply the medication, and then a 15 min debrief on any side effects and comments on the efficacy and feasibility of self-administering the medication. To prevent motion sickness, participants will administer the medication at least 30-45 min before the motion starts (e.g., centrifuge, launch, re-entry). To use the medication to treat motion sickness, participants will administer the medication while symptoms are still mild. Following the operational exercise, a short survey will be used to obtain the timing of the administration relative to the motion stressor, the operational environmental conditions (e.g., sea state or centrifugation levels), description of motion sickness symptoms and side effects, and subjective comments about the feasibility and efficacy of intranasal scopolamine gel.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will involve astronauts assigned to spaceflight missions or test personnel assigned to operational activities that involve provocative motion (e.g., simulations or parabolic flights).
2. No participants should have no neurologic, vestibular or autonomic disorders, or medical conditions that could be worsened by scopolamine (narrow-angle glaucoma or urinary retention)
3. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) negative test, confirmed by Food and Drug Administration (FDA) authorized COVID-19 test < 7 days prior to study drug administration or no COVID 19 symptoms up to 10 days prior to study drug administration.

Note: There are no accepted forms of terrestrial motion analogs that adequately predict susceptibility to space motion sickness so none will be used in this field test.

Exclusion Criteria:

1. Subjects will be excluded if they are taking other drugs that are capable of causing CNS effects such as antihistamines, tricyclic antidepressants, and muscle relaxants or have hypersensitivity to scopolamine or other belladonna alkaloids or to any ingredient or component in the formulation or delivery system.
2. Pregnant women are excluded from participation. Women of child-bearing potential will be offered a pregnancy screening test and excluded with a positive test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Motion sickness (MS) symptoms using Pensacola Diagnostic Index (PDI) nausea scale. | 1 week
  The maximum nausea score (from 0 = none to 3 = severe) will be recorded once for each of the first three inflight days and once for each of the first three postflight days, or once per operational setting not involving spaceflight (e.g., once per simulation or parabolic flight).

SECONDARY OUTCOMES:
Motion sickness symptom severity using a Subjective Discomfort Rating (SDR). | 1 week
  The SDR scale ranges from 0-20 with higher numbers reflecting greater symptom severity (20 = vomiting).
Vertigo severity | 1 week
  Vertigo severity on a score (from 0 = none to 3 = severe) will be obtained once for each of the first three inflight days and once for each of the first three postflight days when space motion sickness is present, or once per operational setting not involving spaceflight (e.g., once per simulation or parabolic flight).
Headache severity | 1 week
  Headache severity on a score (from 0 = none to 3 = severe) will be obtained once for each of the first three inflight days and once for each of the first three postflight days when space motion sickness is present, or once per operational setting not involving spaceflight (e.g., once per simulation or parabolic flight).
Drowsiness severity | 1 week
  Drowsiness severity on a score (from 0 = none to 3 = severe) will be obtained once for each of the first three inflight days and once for each of the first three postflight days when space motion sickness is present, or once per operational setting not involving spaceflight (e.g., once per simulation or parabolic flight).
Motion sickness impact on performance of functional tasks (from 0 = none to 4 = severe) | 1 week
  Subjective rating of motion sickness impacts to performance of functional tasks (from 0 = none to 4 = severe) will be obtained once for each of the first three inflight days and once for each of the first three postflight days when space motion sickness is present, or once per operational setting not involving spaceflight (e.g., once per simulation or parabolic flight).

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Wood, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- NASA Johnson Space Center Neuroscience Laboratory, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No